CLINICAL TRIAL: NCT05301803
Title: A Prospective, Single-Center, Open-Label, Single-Arm Study to Evaluate the Safety and Technical Performance of the CathVision ECGenius® System.
Brief Title: An Evaluation of the Safety and Performance of the CathVision ECGenius® System.
Status: Completed | Type: Observational
Sponsor: CathVision ApS (Industry)
Collaborators: Medicept Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-00003-A
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrhythmia
Keywords: electrophysiology; atrial fibrillation; cardiac ablation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrophysiology procedure — Electrophysiology testing and cardiac ablation of arrhythmia

SUMMARY:
The primary objective is to evaluate the safety and technical performance of the CathVision ECGenius® System. The secondary objective is to benchmark the intracardiac electrogram signal quality compared to commercially available systems in patients undergoing assessment and ablation of cardiac arrhythmias.

DETAILED DESCRIPTION:
A prospective, single center, open-label, single arm study to evaluate the safety and technical performance of the CathVision ECGenius® system.

Patients undergoing assessment and ablation of cardiac arrhythmias during an electrophysiology (EP) procedure, and who meet all inclusion criteria will be enrolled in the study and undergo the EP procedure. Intracardiac signals will be passively recorded using the CathVision ECGenius® System in parallel with a commercial EP recording system and later compared and evaluated. The investigational device will not be used for direct clinical care decisions or therapy. The EP procedure will be guided by the study site Standards Of Care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for catheter ablation or diagnostic electrophysiology procedure.
* At least 18 years of age.
* Able and willing to provide informed consent or obtain consent from a legally authorized representative (LAR).

Exclusion Criteria:

* Patient inability to understand or refusal to sign informed consent.
* Patient is a prisoner or under incarceration
* Patients who in the opinion of the physician are not candidates for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients indicated for EP study or cardiac ablation.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel C Thompson, MD PhD, Principal Investigator — The University of Vermont Medical Center
Locations (1):
- The University of vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Consecutive patients referred for an electrophysiology study or cardiac ablation.
Period: Overall Study
Arm/Group | Single Arm
Started | 27
Completed | 25
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.67 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Baseline Noise Comparison
Description: Measure the peak to peak baseline noise in two EP recording systems for both bipolar and unipolar electrograms in μV
Time Frame: EP and ablation procedures can take up to six hours
Population: Baseline noise
Measure: Median (Inter-Quartile Range); unit: μV
Arm/Group | Single Arm
Number analyzed (Participants) | 25
μV
  ECGenius Bipolar Baseline Noise | 19 [11 to 29]
  ECGenius Unipolar Baseline Noise | 46 [20 to 126]
  LabSystem Pro Bipolar Baseline Noise | 31 [22 to 38]
  LabSystem Pro Unipolar Noise | 463 [138 to 525]

2. Primary Outcome: Freedom From Major Adverse Events, Evaluated at Hospital Discharge
Description: Freedom from major adverse events, evaluated at hospital discharge
  Adverse events were categorized as one of:
  An adverse event (AE) A serious adverse event (SAE) An Adverse device effect (ADE) is an AE related to the use of an investigational medical device.
  A Serious adverse device effect (SADE) is an ADE that that has resulted in any of the consequences characteristic of an SAE.
  An unanticipated adverse device effect (UADE) is defined as any serious adverse effect on health, safety, any life-threatening problem, death caused by or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in predicate devices, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.
Time Frame: From EP procedure to discharge is usually one day.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 27
Participants | 26

ADVERSE EVENTS:
Time Frame: from hospital admission to discharge, typically one day.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=27)
Pericardial effusion (Cardiac disorders) | 1 (1) — pericardial effusion after transeptal puncture requiring pericardial drainage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05301803/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT05301803/SAP_001.pdf